CLINICAL TRIAL: NCT01287702
Title: The Impact of Early Feeding Following Ligation of the Acute Bleeding Varices
Brief Title: Early Feeding Following Ligation of Acute Bleeding Varices
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: IRB, E-DA hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: early feeding after ligation
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Varices
Keywords: early feeding; varices bleeding; to evaluate impact of early feeding on early rebleeding after ligation of varices
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early feeding (Experimental): patients receiving EVL will receive liquid diet since 4 hours after arresting of variceal bleedingpatients with acute bleeding varices arrested by EVL
  Interventions: Dietary Supplement: Early feeding
- Dealyed feeding (Active Comparator): patients with acute bleeding varices arrested by EVL, will receive feeding 48 hours after EVL.
  Interventions: Dietary Supplement: Delayed feeding; Dietary Supplement: Dealyed feeding

INTERVENTIONS:
Dietary Supplement: Delayed feeding — patients with acute bleeding varices arrested by EVL, will receive feeding 48 hours after EVL
  Arms: Dealyed feeding
Dietary Supplement: Dealyed feeding — patients with acute bleeding varices arrested by EVL, will receive feeding 48 hours after EVL
  Arms: Dealyed feeding
Dietary Supplement: Early feeding — patients receiving EVL will receive liquid diet since 4 hours after arresting of variceal bleedingpatients with acute bleeding varices arrested by EVL
  Arms: Early feeding

SUMMARY:
The impact of feeding after endoscopic treatment of gastroesophageal varices has never been investigated. It is still unknown whether early feeding may increase early rebleeding in patients with acute esophageal variceal bleeding treated with EVL. It is customary for clinicians to institute fasting for 2 or 3 days after emergency EVL. This may be a safe approach to watch against early rebleeding. However, many patients would be fasting for a longer time and nutrition may be impaired, possibly resulting in aggravation of ascites. Thus, the investigators conduct a controlled study to evaluate whether early feeding have a bad impact on patients receiving emergency EVL or histoacryl injection for bleeding gastric varices.

DETAILED DESCRIPTION:
Acute esophageal variceal hemorrhage is a dreadful complication of portal hypertension. Its management evolved rapidly in recent years. Traditional managements include vasoconstrictor and balloon tamponade. Vasoconstrictors have been shown to control approximately 80% of bleeding episodes, are generally used as a first line therapy. Following the use of vasoconstrictor, endoscopic therapy is often employed to arrest the bleeding varices as well as preventing early rebleeding. Meta-analysis showed that the combination of vasoconstrictor and endoscopic therapy is superior to endoscopic therapy alone in the control of acute esophageal variceal hemorrhage. Our previous study showed that endoscopic variceal ligation (EVL) is superior to Endoscopic injection sclerotherapy (EIS) in the control of active variceal hemorrhage. It is thus recommended that EVL is the first enscopic treatment of choice for acute esophageal variceal bleeding. Moreover, apart from the control of acute variceal bleeding, prophylactic antibiotics has been proven to be helpful in the prevention of bacterial infection as well as preventing early variceal bleeding. With the advent of new treatment modalities and measures taken to approach patients with acute esophageal variceal bleeding, the mortality of acute esophageal variceal bleeding is significantly reduced in recent years.

On the other hand, early rebleeding due to ligation-induced ulcer may be encountered. The impact of feeding after endoscopic treatment of gastroesophageal varices has never been investigated. It is still unknown whether early feeding may increase early rebleeding in patients with acute esophageal variceal bleeding treated with EVL. It is customary for clinicians to institute fasting for 2 or 3 days after emergency EVL. This may be a safe approach to watch against early rebleeding. However, many patients would be fasting for a longer time and nutrition may be impaired, possibly resulting in aggravation of ascites. Thus, we conduct a controlled study to evaluate whether early feeding have a bad impact on patients receiving emergency EVL or histoacryl injection for bleeding gastric varices.

Methods of treatment:

Enrolled Criteria:

1. The etiology of portal hypertension is cirrhosis.
2. Age ranges between 20-80 y/o.
3. Patients presenting with acute gastroesophageal variceal bleeding proven by emergency endoscopy within 12 hours. (Acute esophageal variceal bleeding was defined as: 1) when blood was directly seen by endoscopy to issue from an esophageal varix (active bleeding), or 2) when patients presented with red color signs on their esophageal varices with blood in esophagus or stomach and no other potential site of bleeding identified (inactive bleeding). Gastric variceal bleeding is defined as active spurting from a gastric varix or presence of red spots on a gastric varix.
4. EVL is performed after confirmation of acute esophageal variceal bleeding. Histoacryl injection is performed if acute gastric variceal bleeding is diagnosed. Bleeding is arrested on the spot.

Exclusion criteria:

1) association with severe systemic illness, such as sepsis, COPD, uremia, HCC, > BCLC stage B 3)failure in the control of bleeding by emergency endoscopic treatment. 4)moribund patients, died within 12 hours of enrollment 5)Uncooperative 6) Ever received EIS, EVL within one month prior to index bleeding 7)Child-Pugh's scores > 13 8) Deep jaundice (serum bilirubin > 10 mg/dl), presence of encephalopathy > stage II or massive ascites

Eligible subjects will receive vasoconstrictor for 3 days (either terlipressin or somatostatin), prophylactic antibiotics for 5 days (cephazolin or norfloxacin 400mg bid), lactulose. Eligible subjects will be randomized to 2 groups. Group 1 will be allowed to take liquid diet (fruit juice, soy bean juice, milk, rice in liquid form) for 3 days within 4 hours after endoscopic treatment. Additionally, intravenous fluid less than 500 cc per day will be given. Subsequently, soft diet will be given for 4 days, and on regular diet on the 8th day after endoscopic treatment.

Group 2 will be fasting for 48 hours after endoscopic treatment and intravenous fluids (normal saline or glucose water) 1500 cc per day with electrolytes will be administered for 2 days. After 2 days of fasting, if rebleeding does not occur, liquid diet will be given for one day, subsequently, soft diet for 4 days, and on regular diet on the 8th day after endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The etiology of portal hypertension is cirrhosis.
2. Age ranges between 20-80 y/o.
3. Patients presenting with acute gastroesophageal variceal bleeding proven by emergency endoscopy within 12 hours. (Acute esophageal variceal bleeding was defined as: 1) when blood was directly seen by endoscopy to issue from an esophageal varix (active bleeding), or 2) when patients presented with red color signs on their esophageal varices with blood in esophagus or stomach and no other potential site of bleeding identified (inactive bleeding). Gastric variceal bleeding is defined as active spurting from a gastric varix or presence of red spots on a gastric varix.
4. EVL is performed after confirmation of acute esophageal variceal bleeding. Histoacryl injection is performed if acute gastric variceal bleeding is diagnosed. Bleeding is arrested on the spot.

Exclusion Criteria:

1. association with severe systemic illness, such as sepsis, COPD, uremia, HCC, > BCLC stage B
2. failure in the control of bleeding by emergency endoscopic treatment.
3. moribund patients, died within 12 hours of enrollment
4. Uncooperative
5. Ever received EIS, EVL within one month prior to index bleeding
6. Child-Pugh's scores > 13
7. Deep jaundice (serum bilirubin > 10 mg/dl), presence of encephalopathy > stage II or massive ascites

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Success rate of initial hemostasis | 48 hours
  hemostasis for 48 hours after ligation
very early rebleeding rate | 48- 120 hours
  rebleeding during this period
ulcer bleeding rate | 14 days
  14 days after ligation of varices

SECONDARY OUTCOMES:
The amount of blood transfuion and mortality | 14 days
  The amount of blood transfuion and mortality with 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan